CLINICAL TRIAL: NCT05608629
Title: Vagus Nerve Stimulation as Treatment for Long Covid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Benjamin Natelson, Professor of Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01846
Record Dates: First submitted 2022-11-04; First posted 2022-11-08 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Long COVID; Chronic Fatigue Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Application of electrode to left tragus with stimulus intensity at that which is just below pain threshold for 35 min a day for 6 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcutaneous Non-Invasive Vagus Nerve Stimulation (Experimental): Application of electrode to left tragus with stimulus intensity at that which is just below pain threshold for 35 min a day
  Interventions: Device: Transcutaneous Non-Invasive Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Non-Invasive Vagus Nerve Stimulation — The parasym is a system for delivering a fixed signal to stimulate the auricular branch of the vagus nerve. The device used is available without prescription in UK and EU. Similar devices have been used to treat migraine and one is in testing to be used for atrial fibrillation.

SUMMARY:
Many patients do not recover following Covid infection. The resulting illness is called Long Covid. Because there is no agreed upon treatment for this ailment, the research team has decided to do an open label pilot study using non-invasive, transcutaneous stimulation of the auricular branch of the vagus nerve. Inclusion criteria required the patient to fulfill criteria for having chronic fatigue syndrome. To date, fourteen patients provided evaluable data. Eight of these fulfilled the study's requirements for treatment success.

DETAILED DESCRIPTION:
Patients who have had COVID and who fulfill criteria for chronic fatigue syndrome will sign IC and be mailed a parasym device with instructions its use after completing entry baseline questionnaires. Subjects will be called two, four and six weeks after beginning participation [application of electrode to left tragus with stimulus intensity at that which is just below pain threshold for 35 min a day] to ask about adverse events. At the end of 6 weeks, patients will complete these questionnaires again plus one assessing their assessment of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to have had COVID
* Patients have to fulfill the 1994 case definition for chronic fatigue syndrome.

Exclusion Criteria:

* BMI > 30

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Natelson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to benjamin.natelson@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be determined.)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous Non-Invasive Vagus Nerve Stimulation
Started | 17
Completed | 15
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Transcutaneous Non-Invasive Vagus Nerve Stimulation
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: Treatment success is defined as patient had to improve on 2 of the following:
  a 14% improvement in SF-36 -- physical function (0-100 scale, higher score = less disability;
  report of marked or moderate improvement (2-3 on a scale going from +3 to -3] based on the treatment [patient global indication of change (0-7, higher score = more improvement);
  going from fatigue case to no fatigue on Chalder fatigue scale (0-3, higher score = more fatigue;
  improvement on VAS of at least 2 points [VAS going from none [0] to 5 [very severe] with at least a 3 [substantial] on one of the following Sx --> fatigue, brain fog, widespread pain
Time Frame: Baseline to post-treatment at 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Non-Invasive Vagus Nerve Stimulation
Number analyzed (Participants) | 15
Participants | 8

2. Secondary Outcome: Number of Participants With Change in the Profile of Mood States (POMS)
Description: Number of participants with reductions of at least 10 points on the short version of the Profile of Mood States. The POMS ranges from 0 -120. Higher score indicates poorer health outcomes.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Non-Invasive Vagus Nerve Stimulation
Number analyzed (Participants) | 15
Participants | 5

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Transcutaneous Non-Invasive Vagus Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT05608629/Prot_000.pdf